CLINICAL TRIAL: NCT00597025
Title: Impact of Providing High Protein Bar to Dialysis Patients With Low Serum Albumin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Satellite Healthcare (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SR017PB
Record Dates: First submitted 2008-01-08; First posted 2008-01-17 (Estimated); Last update posted 2020-03-20 (Actual); Status verified 2019-04

CONDITIONS: End Stage Renal Disease; Hypoalbuminemia; Malnutrition
Keywords: Malnutrition; Hypoalbuminemia; Dietary Supplements; Hemodialysis; Peritoneal Dialysis
MeSH Terms: conditions — Kidney Failure, Chronic; Hypoalbuminemia; Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Group A (Active Comparator): Center Hemodialysis patients
  Interventions: Dietary Supplement: Protein Food Bar Intelligent Indulgence
- Group B (Active Comparator): Center hemodialysis patients
  Interventions: Dietary Supplement: Protein Food Bar Intelligent Indulgence
- Group C (No Intervention): Center Hemodialysis Patients
- Group D (Active Comparator): Peritoneal dialysis patients
  Interventions: Dietary Supplement: Protein Food Bar Intelligent Indulgence
- Group E (No Intervention): Peritoneal dialysis patients

INTERVENTIONS:
Dietary Supplement: Protein Food Bar Intelligent Indulgence — Patients will be given one protein bar at each dialysis treatment, 3 times per week for 3 months
  Arms: Group A
Dietary Supplement: Protein Food Bar Intelligent Indulgence — Patients will be given 7 bars per week. In addition to the the three bars given on Hemodialysis each week, the patients will be given on the first treatment of the week four protein bars to be eaten on non-dialysis days
  Arms: Group B
Dietary Supplement: Protein Food Bar Intelligent Indulgence — Patients will be given a monthly supply of protein bars to provide for daily intake of one protein bar.
  Arms: Group D

SUMMARY:
This study is to evaluate the impact of providing high protein supplementation in the form of a medical food bar containing 20grams of protein eath to hypoalbuminemic dialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with ESRD undergoing center hemodialysis or peritoneal dialysis for more than 90 days.
* 18 years of age or older.
* Must have a reasonable expectation of remaining on treatment for at least 3 months.
* Must have an average serum albumin of <3.5 g/dL over the three months prior to entry into the study.
* Must be able to understand and sign the informed consent.
* Must be willing and able to participate in nutrition interviews for determination of nutrient intake from conventional foods.

Exclusion Criteria:

* Allergy to protein, milk, nuts or wheat.
* Documented ongoing acute infection or inflammatory process including treatment with antibiotics within a two week time of study entry.
* Severe acidosis defined as pre-dialysis serum bicarbonate levels of <15 mEq/L.
* Presence of conditions that would affect normal response to repletion of protein and calories, such as gastrointestinal disorders including inflammatory bowel disease.
* Hospitalization for an infectious condition within 4 weeks prior to study entry.
* Planned surgery within the three month study period including planned kidney transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 375 (Estimated)
Dates: Start 2007-12 (Actual); Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
The mean change (from baseline to month 3) in serum albumin levels among study groups and the proportion of patients treated with the protein food bar reaching an increase of 0.3 g/dL over the three month study period. | Each month for the three months.
Incidence of potential adverse events including nausea, vomiting, diarrhea, acidosis, and uremic symptoms as evidenced by clinical symptoms and possible worsening of laboratory measures such as BUN, Kt/V, nPNA and bicarbonate. | Each month for 3 months

SECONDARY OUTCOMES:
Proportion of patients who reached the goal albumin of >3.5 g/dL during the study period | Month 3
Overall acceptance and compliance of bar form medical food over a 3 month period will be assessed via the proportion of patients who ingested 75% or more of the recommended bars. | Each month for 3 months
Impact of protein intake on laboratory measures such as pre-albumin, CRP and ferritin will be monitored | Each month for 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte Schiller-Moran, MD, Principal Investigator — Satellite Healthcare, Inc.
Locations (2):
- United States (2):
  - Satellite Healthcare, Inc., Mountain View, California
  - WellBound, Inc., Mountain View, California